CLINICAL TRIAL: NCT06230900
Title: Assessment of Mass Balance of Orally Administered [14C] (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one in Healthy Volunteers Using a Microtracer Approach
Brief Title: Mass Balance of Orally Administered [14C] (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one
Acronym: TrueCal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: TNO (Other); Bonumose, Inc. (Unknown); Gelderse Vallei Hospital (Other)
Responsible Party: Principal Investigator, Marlou Dirks, Assistant Professor, Wageningen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL84060.028.23
Record Dates: First submitted 2024-01-07; First posted 2024-01-30 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Energy Intake; Energy Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): 14C (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one ingestion (test period)
  Interventions: Other: (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one; Combination Product: 14C-(3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one

INTERVENTIONS:
Other: (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one — (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one ingestion
Combination Product: 14C-(3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one — 14C (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one ingestion

SUMMARY:
Worldwide almost 40% of the adult population is overweight (including >10% obese), and more than 350 million children (up to the age of 19) are overweight. Overweight and obesity are significant problems and important risk factors for several lifestyle-related diseases, such as cardiovascular disease, certain cancers, non-alcoholic fatty liver disease (NAFLD) and type 2 diabetes (T2D). Excessive consumption of glucose/sucrose is a major contributor to overweight and obesity. Alternative, low-calorie sweeteners could reduce daily energy intake and thus slow down the development of these conditions and related diseases. (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one is a sweetener that may be suitable for use as a sugar substitute; it is only partially digested in the small intestine and as a result has a lower energy density than more traditional sweeteners such as sucrose. However, it is not yet known to what extent (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one is used in the body and then excreted.

The aim of this study is to measure the metabolic utilization (the 'mass balance') of a single dose of 14C-labelled (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one and AMS technology. Based on clinical data of excretion (urine and faeces) and CO2 production (expired air), the mass balance can be derived. These generated results will be used to map the metabolic pathways (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one undergoes during the digestion process. In addition, it will provide insight into the use of AMS technology to investigate the relationship between diet and health.

DETAILED DESCRIPTION:
Objective: To determine the mass balance of (3S,4S,5R)-1,3,4,5,6-Pentahydroxy-hexan-2-one (low GI sweetener) in healthy volunteers.

Study design: Single centre, open-label, non-randomised, single oral administration study Study population: 8 healthy males and females (18-65 y, BMI 18.5-25 kg·m-2) Intervention: Orally ingestion of 14C-labelled (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one, followed by a 72-hour test period during which all urine and faeces will be collected, as well as repeated sampling of blood and expired air, as well as indirect calorimetry measurements.

Main study parameters/endpoints: Mass balance of (3S,4S,5R)-1,3,4,5,6-Pentahydroxy-hexan-2-one following 14C-(3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one ingestion. Secondary endpoints: content of 14C-labelled metabolites in carbohydrate metabolism pathways, routes of elimination of (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one. Ventilated hood measurements will be used as proof of concept to assess caloric value of carbohydrates.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Insertion of the catheters in a vein is comparable to a normal blood draw and the only risk is a small local hematoma. (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one ingestion might lead to gastro-intestinal discomfort. During the adaptation period participants will consume food-grade (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one, which is safe for human consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females using contraception during and for 3 months after the study, aged from 18-65 years at the time of signing the informed consent
* 18.5<BMI<25kg.m2
* Willing and able to communicate and participate in the whole study, including consumption of (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one and meals offered during study conduct
* Regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)
* Usually eat 3 meals per day (i.e. breakfast, lunch and dinner)

Exclusion Criteria:

* Any diagnosed metabolic Impairment (e.g. Type 1 or 2 diabetes)
* Any diagnosed cardiovascular disease
* Hypertension (≥140 mmHg systolic and/or ≥90 mmHg diastolic)
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastro-intestinal disease, immunodeficiency, endocrine, neurological or psychiatric disorders
* Any diagnosed respiratory disease, such as COPD or asthma
* Any previous motor disorders or disorders in muscle and/or lipid metabolism
* Known severe kidney problems
* Presence of an ulcer in the stomach or gut and/or strong history of indigestion
* Recent or chronic history of diarrhoea
* Known anaemia
* A personal or family history of thrombosis (clots), epilepsy, seizures, or schizophrenia.
* Regular use of dietary supplements (>3 times per week)
* Chronic use of any prescribed or over the counter pharmaceuticals (excluding oral contraceptives and contraceptive devices)
* History of any drug or alcohol abuse in the past two years
* Drug use
* Claustrophobia
* On a weight loss diet (including intermittent fasting) or following a high calorific/high protein diet in order to gain weight
* Functional constipation
* Any known food allergies or intolerances to the 14 major food allergens (celery, cereals containing gluten, crustaceans, eggs, fish, lupin, milk, molluscs, mustard, tree nuts, peanuts, sesame seeds, soybeans, sulphur dioxide and sulphites) or history of a malabsorption syndrome including coeliac disease
* Regular gastrointestinal complaints including abdominal pain, stomach upsets and borborygmi or known or suspected irritable bowel syndrome
* Currently taking part in other scientific research
* Received a product with 14C in the past 12 months
* Pregnant or breastfeeding
* Smoking or having used nicotine-containing products in the 6 months prior to the study.
* Taken antibiotics within the 60 days prior to the adaptation period.
* Currently involved in a structured progressive resistance training programme (>3 times per week)
* Sedentary lifestyle as assessed using the International Physical Activity Questionnaire [IPAQ].
* Employed or undertaking a thesis or internship at the department of Human and Animal Physiology or TNO (department of Metabolic Health Research)
* Unable to give consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
14C (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one mass balance | day 0-3 test period
  Mass balance recovery after a single oral dose of 14C (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one

SECONDARY OUTCOMES:
14C (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one elimination routes | day 0-3 test period
  Mass balance recovery after a single oral dose of 14C (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one
Metabolite profiling of (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one metabolites | day 0-3 test period
  Plasma, urine and faecal metabolite profiling of (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one metabolites
Quantification of (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one metabolites | day 0-3 test period
  Plasma, urine and faecal quantification of (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one metabolites
Structural identification of (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one metabolites | day 0-3 test period
  Plasma, urine and faecal structural identification of (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one metabolites
Resting energy expenditure | day 0-3 test period
  REE based on the Weir formula
(3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one pathway activity | day 0-3 test period
  (3S,4S,5R)-1,3,4,5,6-pentahydroxy-hexan-2-one pathway activity
Rate of whole-body substrate oxidation | day 0-3 test period
  Rate of whole-body substrate oxidation (i.e. carbohydrate and lipid oxidation) measured via indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Marlou Dirks, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands